CLINICAL TRIAL: NCT03842527
Title: Pre-Operative Gastric Volume Assessment Following Carbohydrate-Loading in Obstetrical Patients Undergoing Elective Cesarean Section: A Randomized Clinical Pilot Study
Brief Title: Gastric Voume Assessment for Aspiration Risk in OB ERAS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Heather Hurdle, Anesthesiologist, Clinical Assistant Professor, Department of Anesthesiology, Perioperative and Pain Medicine, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: REB17-2345
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Cesarean Section
Keywords: Gastric Ultrasound; Carbohydrate Loading
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Fasting Group (Active Comparator): Ultrasound scan of gastric antrum 1 hour prior to procedure. Patients assigned to this group will follow standard fasting procedures of no eating or drinking 8 hours prior to C-section.
  Interventions: Device: Ultrasound
- Carbohydrate Loading Group (Experimental): Ultrasound scan of gastric antrum 1 hour prior to procedure.
  Patients assigned to this group must stop eating 8 hours prior to their scheduled C-section time.
  The night before their C-section they must drink 800mL of 100% apple juice (not from concentrate) OR 800mL of cranberry juice cocktail, not both
  The day of their C-section, starting 3 hours before surgery and to be finished 2 hours before surgery time, patients must drink 400mL of 100% apple juice OR 400mL of cranberry juice cocktail, not both
  Please note:
  * The apple juice must be 100% juice, not from concentrate
  * The cranberry juice cocktail must not be plain cranberry juice
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Gastric ultrasound of the stomach antrum to assess contents 1 hour prior to C-section surgery. Scans will be completed in both supine (lying on back) and right lateral decubitus (positions) positions. The completion of both scans will take 5-10 minutes total

SUMMARY:
In recent years, human and animal studies have found that carbohydrate-loading prior to surgery leads to improved response to surgical stress and improved postoperative well-being when compared to traditional fasting guidelines. Such positive findings have lead to the increased use of preoperative intake of carbohydrate rich drinks prior to elective surgeries.

However, one of the biggest risks during surgery when a patient is asleep is having stomach contents come up into the lungs. For this reason, a stomach that is empty or has minimal amount of contents is safest. Historically, patients have been instructed not to eat or drink for 8 hours before surgery because it was thought to lower the risk of having fluid or contents in the stomach. This is the current practice patients are asked to follow before undergoing a C-section. However, non-pregnant patients undergoing other surgeries are instructed to have carbohydrate-rich drinks because of the potential benefits. Using ultrasound, the abdomen can be simply scanned to see if there are stomach contents present before surgery. This can allow for the potential determination of what the aspiration risk may be.

What the investigators want to do is look at the safety of using carbohydrate-loading in patients having a C-section. The investigators want to make sure that patients who follow carbohydrate-loading by having a clear, sugary drink 3 hours before a C-section are not at greater risk of having a large amount of stomach contents and be at higher risk of aspirating. This will be done by taking an ultrasound scan of the stomach that will tell the investigators if there are contents in the stomach and whether there is a risk of aspiration.

Patients having an elective C-section will be randomized into two groups. The first group will follow carbohydrate-loading by having a drink of apple juice or cranberry juice cocktail the night before (800mL) and 3 hours before (400mL) the C-section. The second group will follow standard practice of not eating or drinking less than 8 hours prior to surgery. An anesthesiologist will ultrasound the stomach 1 hour before the scheduled procedure time. The first ultrasound will be completed in the supine position (lying on back). The second will be done in the right lateral decubitus position (lying on right side). This should not take more than 5-10 minutes total.

ELIGIBILITY:
Inclusion Criteria:

* Non-laboring pregnant women
* ≥36 weeks gestational age
* scheduled elective cesarean delivery
* ≥18 years of age
* ASA physical status I to III
* weight 50 to 120 kg
* height ≥150 cm
* Ability to understand the rationale of the study assessments

Exclusion Criteria:

* multiple gestation
* abnormal anatomy of the upper gastrointestinal tract
* gestational diabetes or pre-existing diabetes mellitus
* previous surgical procedures on the esophagus, stomach, or upper abdomen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade 2 antrum | 1 hour prior to C-section delivery
  Clear fluid is evident in antrum in both supine and right lateral decubitus scanning positions

SECONDARY OUTCOMES:
Incidence of Grade 0 antrum | 1 hour prior to C-section
  Antrum appears empty in both supine and right lateral decubitus scanning positions
Incidence of Grade 1 antrum | 1 hour prior to C-section
  Antrum appears empty in supine position, but clear fluid is visible in right lateral decubitus position
Cross-sectional antral area | 1 hour prior to C-section
  Cross-sectional area measurement of the gastric antrum

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta